CLINICAL TRIAL: NCT03169946
Title: Effects of Chlorhexidine-Metronidazole Combination as an Intracanal Medicament on Periodontal Healing in Concurrent Endodontic Periodontal Lesions With Communication: A Randomized Controlled Clinical Study
Brief Title: Chlorhexidine-Metronidazole Combination as an Intracanal Medicament on Periodontal Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: kirtika perio 2015
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Periodontal and Endodontic Lesion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Active Comparator): Endodontic treatment using chlorhexidine metronidazole combination as an intracanal medicament along with open flap debridement (RCT with CHX-MTZ,OFD).
  Interventions: Procedure: RCT with CHX-MTZ,OFD
- Positive Control Group : (Active Comparator): Endodontic treatment using chlorhexidine as an intracanal medicament along with surgical periodontal therapy in form of open flap debridement(RCT with CHX,OFD).
  Interventions: Procedure: RCT with CHX,OFD

INTERVENTIONS:
Procedure: RCT with CHX-MTZ,OFD — Endodontic treatment using chlorhexidine metronidazole combination as an intracanal medicament along with open flap debridement .
  Arms: Test Group
Procedure: RCT with CHX,OFD — Endodontic treatment using chlorhexidine as an intracanal medicament along with surgical periodontal therapy in form of open flap debridement.
  Arms: Positive Control Group :

SUMMARY:
Considering the beneficiary properties of both Chlorhexidine (CHX) and Metronidazole (MTZ) such as property of substantivity and diffusion of these drugs on the external surfaces through the anatomical communication channels in between the root canals and periodontium, may be utilized as an alternative approach for the delivery of drug ( intracanal medicament) in the deep periodontal pockets in concurrent endodontic- periodontic lesion with communication lesions. Thus the aim of study is to conduct a prospective randomized controlled clinical trial to evaluate and compare the effects of CHX-MTZ combination with chlorhexidine alone as an intracanal medicament on periodontal healing in concurrent endodontic- periodontic lesion with communication.

DETAILED DESCRIPTION:
INTRODUCTION

The pulp tissue within the tooth and surrounding periodontium are interrelated to each other due to structural, functional and microbiological similarities. Cross infection of bacterial colonies take place in between these sites through dentinal tubules, apical foramen, lateral and accessory canals.Concurrent endodontic- periodontic lesions are those lesions where both endodontic and periodontal diseases occurring at same time in relation to single tooth.

Endodontic infection present in tooth is responsible for more bone loss, attachment loss and results in impaired healing of periodontium and vice versa.

Complete elimination of microorganisms from infected root canal is very challenging and complicated task. It has been reported that bacteria may survive within the root canal even after chemomechanical preparation, these remaining bacteria again multiply within the root canal. So, intracanal medicament is used as an adjunct to mechanical preparation in disinfection of root canal system.

Chlorhexidine (CHX) is widely used as an intracanal medicament because of its high antimicrobial action, against gram positive and gram negative bacteria.

Antibacterial substantivity of CHX is significantly higher than other medicaments. Various microbiological studies found the reduction in bacterial adherence, lager zones of microbial inhibition after application of CHX as an intracanal medicament. Raheja et al described that 2% CHX gel as an intracanal medicament provide substantive antibacterial activity for sufficiently long periods of time and helps in better healing of endodontic periodontal lesions without communication in their clinical study. Although, CHX is very effective as an intracanal medicament, but can't be used as an final irrigant due to it allergic, hypersensitive reaction, precipitation formation with sodium hypochlorite, EDTA, saline and ethanol and its inability to dissolve necrotic tissue.

In endodontic and periodontal treatment, antibiotics are valuable adjunctive for management of bacterial infections. Local application of antibiotics is considered more effective than systemic administration because of potential risk of adverse effects associated with systemic application.Metronidazole(MTZ) is nitroimidazole compound having broad antibacterial spectrum of bactericidal action mainly against anaerobic microorganisms. MTZ is given along with ciprofloxacin and minocycline as a combination in 3M antibiotic paste in the form of intracanal medicament. Kargul et al in a clinical study showed that there was no abscess formation and pathologic mobility when metronidazole is used as an intracanal medicament.Observations based on in vitro study showed that MTZ-CHX combination was better than calcium hydroxide as an intracanal medicament against E.faecalis.

Keeping in mind the above observations and considering the beneficiary properties of both CHX and MTZ such as property of substantivity and diffusion of these drugs on the external surfaces through the anatomical communication channels in between the root canals and periodontium, may be utilized as an alternative approach for the delivery of drug ( intracanal medicament) in the deep periodontal pockets in these lesions. Thus the aim of study is to conduct a prospective randomized controlled clinical trial to evaluate and compare the effects of CHX-MTZ combination with chlorhexidine alone as an intracanal medicament on periodontal healing in concurrent endodontic- periodontic lesion with communication.

MATERIAL AND METHOD

This study will be conducted in Department of Periodontics and Oral Implantology in collaboration with Department of Conservative Dentistry and Endodontics, Post Graduate Institute of Dental Sciences (PGIDS), Rohtak. The study protocol is according to the ethical standards of Helinski declaration 1975 as revised in 2013.

STUDY POPULATION

Patients will be recruited from regular outpatient department of the periodontics, endodontics and oral medicine PGIDS, Rohtak. The study will be conducted as follows:

Interventional study: This randomized controlled clinical trial will include minimum 36 patients which will be further divided into two groups.

Test Group (n≈ 18)

Treatment involves endodontic treatment using intracanal medicament (chlorhexidine metronidazole combination) along with open flap debridement.

Positive Control Group (n≈ 18)

Treatment involves endodontic treatment using chlorhexidine alone as an intracanal medicament along with surgical periodontal therapy in form of open flap debridement.

METHODOLOGY

Patients will be randomly allocated to control and test groups. The study will be conducted as follows:

1. Presurgical therapy: which will be including

   * Oral hygiene instructions and patient motivation
   * Full mouth supragingival and subgingival scaling and root planning with ultrasonic scaler (EMS Piezon 250, Switzerland), hand scaler and curettes (Hu-Friedy) will be completed in two sessions.
   * Root canal therapy will be initiated in both the groups.
   * In Test group- Metronidazole-chlorhexidine combination (metronidazole-15mg, chlorhexidine gluconate-0.5%w/w)as an intracanal medicament and in positive control group 2% chlorhexidine gel will be placed in root canals. In both groups, total duration for medicament placement will be of 4 weeks.
2. Surgical therapy : After 2 weeks of intracanal medicament placement in both test group and in control group, periodontal surgical procedure in the form of open flap debridement will be performed in both groups.
3. At the time of periodontal surgical procedure, intracanal medicament will be replaced with fresh one and will be remained in the root canals further for 2 weeks (medicament placed for total duration of 4 weeks), after that obturation will be done in both groups.

A probing stent will be fabricated for every patient irrespective of the group, relative to which attachment level, pocket probing depth will be measured.

CLINICAL PARAMETERS

1. Full mouth indices to be recorded at baseline

   * Plaque index(PI)
   * Gingival index(GI)
   * Bleeding on probing(BOP)
   * Probing Pocket depth(PPD)
   * Clinical attachment loss(CAL)
2. Site specific indices

   * Plaque index(PI)
   * Gingival index(GI)
   * Relative Probing Pocket depth(RPPD)
   * Relative Attachment Loss (RAL)
   * Bleeding on probing (BOP)
   * Tooth mobility
   * Relative Gingival Marginal Level (RGML)

Using UNC 15 periodontal probe at 6 sites (mesiobuccal, distobuccal, mesiolingual, distolingual, and median points at buccal and at lingual aspects) per tooth except 3 rd molars for PPD, BOP, GML and CAL while 4 surfaces (mesial, distal, median points at buccal and lingual aspect) will be measured for PI, GI.

Customized bite blocks and parallel angle technique will be used to obtain radiographs.

Clinical parameters will be recorded at baseline, 2 weeks of endodontic treatment and at 3 months, 6 months of periodontal surgery.

PERIODONTAL NON SURGICAL PROCEDURE

This involves supragingival and subgingival scaling and root planing to be performed with ultrasonic scaler, hand scaler and curette and will be completed in minimum two sessions along with patient education and motivation.

ENDODONTIC PROCEDURE

After achieving local anaesthesia, access opening will be made with the help of round bur. Then the root canal will be thoroughly debride followed by copious irrigation and subsequently prepared with the help of endo files. After preparation of the canal, chlorhexidine- metronidazole combination as an intracanal medicament will be placed in test group, chlorhexidine medicament in positive control group and access cavity will be sealed with suitable sealer and medicament left inside for the above mentioned time period. Obturation will be performed with gutta percha and zinc oxide eugenol based sealer.

PERIODONTAL SURGICAL PROCEDURE

After administration of local anaesthesia, buccal and lingual/palatal intracrevicular incision will be made and mucoperiosteal flaps will be reflected including at least one tooth ahead and another behind the tooth. Meticulous defect debridement and root planing will be carried out using area specific curettes and scalers to remove all the granulation tissue. After instrumentation, the root surfaces will be washed with saline solution in attempt to remove any remaining detached fragments from the defect and surgical field. After debridement mucoperiosteal flaps will be repositioned and secured by using 3-0 non absorbable black silk surgical suture. The surgical area will be protected and covered with periodontal dressing and post operative instructions will be given.

POST OPERATIVE CARE

* Suitable antibiotics and analgesics will be prescribed for 5 days.
* Periodontal dressing and sutures will be removed after 1 week.
* Instructions will be given for gentle brushing with soft brush and reinstructed for proper oral hygiene postoperatively and will be examined weekly for up to 1 month after surgery and again at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age between 18-55 years with generalized chronic periodontitis will be enrolled, having at least one tooth with concurrent endodontic periodontal lesion with communication including following features:

  * a clinical and radiographic diagnosis of concurrent endodontic periodontal lesion
  * Wide base pocket, deep probing pocket depth
  * Non vital tooth on the basis of pulp sensibility tests along with periapical radiolucency
  * Radiographic alveolar bone (marginal bone) destruction with apical communication
* Patients of generalized chronic periodontitis will be selected on the basis of Armitage classification of periodontal diseases and conditions [≥30% sites involved with clinical attachment level (CAL) 1-2mm (mild) or 3-4mm (moderate) or ≥5mm (severe)]
* Patients should have more than 20 teeth in their oral cavity excluding third molars.

Exclusion Criteria:

* Systemic illness known to affect the periodontium or outcome of periodontal therapy.
* Patient taking medications such as corticosteroids, calcium channel blockers and anticoagulant therapy, which are known to interfere periodontal wound healing or patient on long term NSAID therapy or bisphosphonates.
* Patients allergic to medication (chlorhexidine, local anaesthetic, antibiotics, NSAID).
* Patients with acute symptoms.
* Pregnant or lactating females.
* Smokers (current and past) and tobacco chewers.
* Grade 3 mobile teeth.
* Unrestorable tooth.
* Root resorption.
* Fractured/perforated roots.
* Developing permanent tooth.
* Abutments.
* Previously root canal filled tooth.
* Patients with aggressive periodontitis
* History of periodontal treatment within 6 months prior to study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-10-14 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
PPD | 6 and half months
  Probing pocket depth
CAL | 6 and half months
  Clinical attachment loss

IPD SHARING:
Plan to Share IPD: Yes